CLINICAL TRIAL: NCT02014727
Title: Safety and Immunogenicity of Recombinant Pichia Pastoris AMA1-DiCo Candidate Malaria Vaccine With GLA-SE and Alhydrogel ® as Adjuvant in Healthy Malaria Non-Exposed European and Malaria Exposed African Adults:a Staggered Phase Ia/Ib, Randomised, Double-blind, Multi-Centre Trial
Brief Title: Safety and Immunogenicity of Recombinant Pichia Pastoris AMA1-DiCo Candidate Malaria Vaccine With GLA-SE and Alhydrogel ® as Adjuvant in Healthy Malaria Non-Exposed European and Malaria Exposed African Adults
Acronym: AMA1-DiCo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: EVI Industries, Inc. (Other); BPRC (Unknown); Recherche Clinique Paris Descartes Necker Cochin Sainte Anne (Other); Centre national de recherche et de formation sur le paludisme (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C12-18 AMA-DiCo; 2013-001920-20 (EudraCT Number)
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2015-09

CONDITIONS: Malaria, Falciparum
Keywords: Malaria vaccine; phase 1,; AMA1-DiCO
MeSH Terms: conditions — Malaria, Falciparum | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AMA1-DiCo + Alhydrogel (Experimental): AMA1-DiCo: 50µg Alhydrogel® : 0.85 mg Al3+ per dose Route : Intramuscular Vaccination schedule : Do, W4, W26
  Interventions: Biological: Group A1 : 50µg AMA1-DiCo + Alhydrogel
- AMA1-DiCo+ GLA-SE (Experimental): Group A2 (15) : European volunteer : AMA1-DiCo + GLA-SE
  AMA1-DiCo: 50µg
  GLA-SE 2.5 µg GLA per dose
  Route : Intramuscular Vaccination schedule : Do, W4, W26
  Interventions: Biological: Group A2 : 50 µg AMA1-DiCo+ GLA-SE
- AMA1-DiCo + GLA-SE (Experimental): Group B1 (18) : African volunteer : AMA1-DiCo + GLA-SE
  AMA1-DiCo: 50µg
  GLA-SE 2.5 µg GLA per dose
  Route : Intramuscular Vaccination schedule : Do, W4, W26
  Interventions: Biological: Group A2 : 50 µg AMA1-DiCo+ GLA-SE
- Placebo (Placebo Comparator): Group B2 (18) : African volunteer : Placebo
  Placebo : isotonic saline solution
  Route : Intramuscular Vaccination schedule : Do, W4, W26
  Interventions: Biological: Group B2 : Placebo

INTERVENTIONS:
Biological: Group A1 : 50µg AMA1-DiCo + Alhydrogel
  Arms: AMA1-DiCo + Alhydrogel
Biological: Group A2 : 50 µg AMA1-DiCo+ GLA-SE
  Arms: AMA1-DiCo + GLA-SE; AMA1-DiCo+ GLA-SE
Biological: Group B2 : Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the safety of 3 doses given at D0, W4, and W26 of 50 µg dosage of AMA1-DiCo adjuvanted either with GLA-SE or Alhydrogel® in healthy European adults not previously exposed to the parasite P.falciparum and in healthy African adults exposed to the parasite. The safety and the tolerability of the vaccine will be assessed on the rate of solicited and unsolicited events/reactions. The safety profile will include local and systemic reactions/events as well as the biological safety, based on a clinically significant change of the baseline value of the main biological criteria.

DETAILED DESCRIPTION:
The project aims are :

-To evaluate the safety of 50 µg AMA1-DiCo malaria vaccine candidate with GLA-SE and Alhydrogel® as adjuvant, in healthy European adults not previously exposed to the parasite Plasmodium falciparum and in healthy African adults exposed to the parasite.

T-o assess the humoral immune response to the vaccine antigens by measuring the level of IgG in all volunteers.

To assess the cellular immune response by measuring the T cell cytokines IL-5 and IFNγ production following in vitro stimulation with the vaccine antigens in all volunteers.

Design :

This trial is a staggered Phase Ia/Ib, Randomised, Double-blind, Multi-center Centre trial.

Two different adjuvants will be assessed, Alhydrogel® and GLA-SE. One dosage of 50 µg/3 injections of AMA1-DiCo will be evaluated for each adjuvant.

Sixty six (66) healthy volunteers will be included into the 2 following cohorts (A and B):

Cohort A: 30 Non-exposed European Volunteers (France) Cohort B: 36 Malaria Exposed African Volunteers (Burkina Faso)

The non-exposed European volunteers (cohort A) will be randomised in a 1:1 ratio into two groups of 15 volunteers per group.

The malaria exposed African volunteers (cohort B) will be randomised in a 1:1 ratio, into two groups of 18 volunteers per group.

European Volunteers: Cohort A (30):

Group A1 (15): 50µg AMA1-DiCo + Alhydrogel® Group A2 (15): 50 µg AMA1-DiCo+ GLA-SE

African Volunteers Cohort B (36) :

Group B1 (18): 50 µg AMA1-DiCo + GLA-SE Group B2 (18): Placebo (isotonic saline solution)

In order to start recruitment in cohort B (Africa), the safety will be evaluated on the data of all European volunteers until Day 7 after 1st immunisation of the last European volunteer Data will be presented to an Independent Data safety Monitoring Board (DSMB) that will be appointed for this trial

ELIGIBILITY:
Inclusion Criteria:

1. Age > 20 and < 45 years healthy female and male
2. General good health based on history and clinical examination.
3. Written informed consent obtained before any trial procedure.
4. Female and male volunteers practicing contraception before and up to four (4) weeks after the third vaccination.
5. Available to participate in follow-up for the duration of trial.
6. Reachable by phone during the whole trial period.
7. Volunteers should be affiliated to a social security regimen

Exclusion Criteria:

1. Positive pregnancy test
2. Active breast feeding
3. Previous participation in any malaria vaccine trial
4. History of blood transfusion within the last 6 months
5. Symptoms, physical signs or laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the trial results or compromise the health of the volunteers.
6. Any clinically significant laboratory abnormalities on screened blood samples outside the normal range, as defined at the clinical trial site.
7. Enrolment in any other clinical trial during the whole trial period
8. Intake of chronic medication, especially immunosuppressive agents (steroids, immunomodulating or immunosuppressive drugs) during the thirteen weeks preceding the screening visit or during the trial period except topical steroid use including intranasal.
9. Any confirmed or suspected immunosuppressive or immunodeficiency condition during the whole trial period
10. Volunteers unable to be closely followed for social, geographic or psychological reasons.
11. Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the trial.
12. History of anaphylaxis or Known severe hypersensitivity to any of the vaccine components (adjuvant or antigen or excipient)
13. Vaccination or gamma globulin: 4 weeks prior and after each vaccination if a vaccination is necessary during this period, the volunteer will be withdrawn from the study.
14. Positive HIV, HBV (Ag HBS) and HCV tests.
15. History of malaria or travel in malaria endemic areas within the past twenty-six weeks.
16. Positive serology for malaria antigen PfAMA-1
17. Intention to travel to malaria endemic countries during the trial period.

    -

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events | Up to four weeks after the third vaccination.
  The safety profile will be assessed in all volunteers on the following criteria:
  * Immediate reactogenicity (reactions within 60 minutes after each vaccination).
  * Local and systemic reactogenicity measured from Day 0 to Week 2 after each vaccination.
  * Any unsolicited adverse event between the first vaccination and four weeks after the third vaccination.
  * Any SAE occurring from the inclusion throughout the trial.

SECONDARY OUTCOMES:
The humoral and cellular responses | 6 months after the last vaccination
  The humoral response to the vaccine antigens (DiCo1, DiCo2 and DiCo3) will be assessed by measuring the level of IgG by ELISA on samples obtained at screening visit Day 0, Week 4, 5, 8, 26, 27, 30 and 52.
  The cellular immune response will be assessed by measuring the T cell cytokine IL-5, and IFNg production by ELISpot following in vitro stimulation with the vaccine antigens on samples obtained at Day 0, Week 26, 30 and 52.

OTHER OUTCOMES:
The quality of the cellular and humoral immune responses | Up to 6 months after the last vaccination
  The quality of the humoral immune response will be assessed by measuring:
  IgG1 and IgG3 subclasses by ELISA on samples obtained at Day 0 and Week 30. IgG responses to four natural allelic variants by ELISA on samples obtained at Days 0 and Week 30.
  An IFA will be employed to verify that the antibodies elicited by the vaccine recognize the native protein on merozoites on samples obtained Day 0 and Week 30.
  Competition ELISA with AMA1 antigen added as competitor at Week 30. The ability to inhibit parasite growth in vitro by a Growth Inhibition Assay (GIA) against at least 3 parasite strains on samples obtained at Day 0, Week 30 and 52.
  IgG avidity by ELISA on a panel of AMA1 alleles at Week 30.
  The quality of the cellular immune response will be assessed by measuring the production of a panel of T cell cytokines in the ELISpot supernatants by multiplex cytokine assay on samples obtained at Day 0, Week 26, 30 and 52.

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, Professor, Principal Investigator — CIC BT505 Cochin Pasteur Groupe Hospitalier Cochin Broca Hotel Dieu. Bâtiment Lavoisier 27, rue du Faubourg Saint-Jacques 75679 PARIS Cedex 14, France odile.launay@cch.aphp.fr; Sodiomon Sirima, Doctor, Principal Investigator — Centre National de Recherche et de Formation sur le Paludisme (CNRFP 01 BP 2208 Ouagadougou 01 1487, Avenue KumdaYonré, Burkina Faso s.sirima.cnlp@fasonet.bf
Locations (2):
- CNRFP, Ouagadougou, Ouagadougou, Burkina Faso
- CIC BT 505 de vaccinologie Cochin Pasteur. Hôpital Cochin Bâtiment Lavoisier 27 rue du faubourg St Jacques., Paris, France

REFERENCES:
- [Result] Sirima SB, Durier C, Kara L, Houard S, Gansane A, Loulergue P, Bahuaud M, Benhamouda N, Nebie I, Faber B, Remarque E, Launay O; AMA1-DiCo Study Group. Safety and immunogenicity of a recombinant Plasmodium falciparum AMA1-DiCo malaria vaccine adjuvanted with GLA-SE or Alhydrogel(R) in European and African adults: A phase 1a/1b, randomized, double-blind multi-centre trial. Vaccine. 2017 Oct 27;35(45):6218-6227. doi: 10.1016/j.vaccine.2017.09.027. Epub 2017 Sep 22. PMID 28947345